CLINICAL TRIAL: NCT04661709
Title: Efficacy and Safety of Chinese Herbal Medicine Wen Xin Granules for the Treatment of Unstable Angina Pectoris With Yang Deficiency and Blood Stasis Syndrome: Study Protocol for a Randomized Controlled Trial
Brief Title: Efficacy and Safety of Wen Xin Granules for the Treatment of Unstable Angina Pectoris
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Collaborators: Special Project of National Traditional Chinese Medicine Clinical Research Base of State Administration of Traditional Chinese Medicine (Unknown); National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Jun Li, Director of cardiovascular department of Guang'anmen Hospital., Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Wenxin granule-20201122
Record Dates: First submitted 2020-11-23; First posted 2020-12-10 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Coronary Heart Disease; Unstable Angina; Chinese Herbal Medicine
Keywords: coronary heart disease; unstable angina; Chinese herbal medicine; Wen Xin granule; traditional Chinese medicine
MeSH Terms: conditions — Coronary Disease; Angina, Unstable | interventions — Clopidogrel; Tablets; Atorvastatin; isosorbide-5-mononitrate; Metoprolol; Trimetazidine; Nitroglycerin

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: It's a double-blind trial and includes two levels of blinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wen Xin granule (Experimental): Patients are given Wen Xin granule by mouth, one dose daily for 2 months & Conventional western medicine, including Aspirin Enteric-coated Tablets 100mg qd, Clopidogrel Hydrogen Sulfate 75 mg qd, Atorvastatin Calcium 20mg qn, Isosorbide Mononitrate Tab 20 mg bid, Metoprolol Tartrate Tab 25mg, Trimetazidine Dihydrochloride Tablets 20mg tid.
  Interventions: Drug: Wen Xin granule; Drug: Clopidogrel Hydrogen Sulfate 75 MG Oral Tablet; Drug: Atorvastatin Calcium; Drug: Isosorbide Mononitrate Tab 20 MG; Drug: Metoprolol Tartrate Tab 25 MG; Drug: Aspirin Enteric-coated Tablets; Drug: Trimetazidine Dihydrochloride Tablets; Drug: glyceryl trinitrate
- WXG placebo (Placebo Comparator): Patients are given Wen Xin granule placebo by mouth, one dose daily for 2 months & Conventional western medicine, including Aspirin Enteric-coated Tablets 100mg qd, Clopidogrel Hydrogen Sulfate 75 mg qd, Atorvastatin Calcium 20mg qn, Isosorbide Mononitrate Tab 20 mg bid, Metoprolol Tartrate Tab 25mg, Trimetazidine Dihydrochloride Tablets 20mg tid.
  Interventions: Drug: Clopidogrel Hydrogen Sulfate 75 MG Oral Tablet; Drug: Atorvastatin Calcium; Drug: Isosorbide Mononitrate Tab 20 MG; Drug: Metoprolol Tartrate Tab 25 MG; Drug: Aspirin Enteric-coated Tablets; Drug: WXG placebo; Drug: Trimetazidine Dihydrochloride Tablets; Drug: glyceryl trinitrate

INTERVENTIONS:
Drug: Wen Xin granule — one dose daily, two times per day.
  Other Names: WXG
  Arms: Wen Xin granule
Drug: Clopidogrel Hydrogen Sulfate 75 MG Oral Tablet — one tablet daily. (for patients who can't use aspirin)
Drug: Atorvastatin Calcium — 20 mg tablet, one tablet each night.
Drug: Isosorbide Mononitrate Tab 20 MG — one tablet， twice daily.
Drug: Metoprolol Tartrate Tab 25 MG — 12.5 mg or 25 mg, two times daily.
Drug: Aspirin Enteric-coated Tablets — 100mg tablet, one tablet daily.
Drug: WXG placebo — one dose daily, two times per day.
  Arms: WXG placebo
Drug: Trimetazidine Dihydrochloride Tablets — 20 mg tablet, one tablet three times daily.
Drug: glyceryl trinitrate — be taken when angina pectoris attacks.

SUMMARY:
This is a double-blind, randomized placebo-controlled trial which aims to evaluate the efficacy and safety of Wen Xin granule in patients with unstable angina pectoris.

DETAILED DESCRIPTION:
Coronary heart disease has remained the leading cause of death worldwide over the past decades. Unstable angina is a clinical syndrome intermediate in severity between stable angina and acute myocardial infarction with high morbidity and mortality. Standard drug therapy and invasive revascularization are effective in decreasing progression to infarction, reducing symptoms and multiple hospitalizations, in most cases without a decrease in the long-term mortality rate. However, there are still many patients with persistence or recurrence of angina despite standard medical therapy and/or revascularization. Wen Xin granule, as a Chinese herbal medicine has shown great effect in patients with unstable angina in our clinical. However, there is still insufficient evidence on his specific efficacy and safety. Therefor, we'd like to evaluate the efficacy and safety of Wen Xin granule in patients with unstable angina through this multi-center, double-blind, randomized placebo-controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* aged between 35 and 75 years of age;
* diagnosed with CAD through coronary arteriography, clinically diagnosed with UAP in low or medium risk;
* belong to Yang deficiency and blood stasis syndrome according to TCM, and give written informed consent.
* For the diagnostic criteria of UAP, the investigators will refer to 2014 AHA/ACC Guidelines for the Diagnosis and Management of Non-ST-Elevation Acute Coronary Syndromes.
* For the TCM diagnostic criteria, the investigators will refer to Guidelines for Clinical Research into New Traditional Chinese Medicine Drugs for Chest Obstruction (2002 edition).

Exclusion Criteria:

* chest pain caused by congenital heart diseases, valvular heart disease, severe neurosis, or arrhythmia
* with New York Heart Association class III or IV heart failure, in acute phase of cerebral infarction;
* with uncontrolled hypertension (systolic blood pressure >160 mmHg and/or diastolic blood pressure >95 mmHg in the resting state)
* with uncontrolled hyperglycemia or diabetic complications, with mental and neurological abnormalities or dysgnosia;
* female patients in pregnancy or lactation;
* by participating in other clinical trials.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 502 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular events | Record the incidence of major adverse cardiovascular events in one year by follow-up.
  Including recurrent angina, acute myocardial infarction, severe arrhythmia, heart failure, and cardiac death.

SECONDARY OUTCOMES:
The thrombelastograph | Before treatment and at eight weeks after treatment.
  Parameters assessed by were R (represent clotting time), K and Angle (reflect clot strength and development), MA (maximum platelet-fibrin clot strength), CI (represents overall coagulability), and LY30 (represents lysis).
TCM symptom scale score | Before treatment, four and eight weeks after treatment.
  TCM syndrome scale includes items of chest tightness, chest pain, heavy body, obesity, phlegm, dark complexion, tongue condition and pulse condition. The chest tightness and chest pain, have 4-grade options of none, mild, moderate and severe, marked as 0, 2, 4 and 6 respectively. The other items have two options of yes or no, marked as 0 and 1 respectively. The higher scores mean more serious symptoms.
Seattle angina questionnaire | Before treatment, four and eight weeks after treatment.
  The SAQ regroups 19 items measuring five specific scales: physical limitations, anginal stability, anginal frequency, treatment satisfaction and disease perception targeting a specific disease and treatment group. Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Li, M.D., Study Director — Guang'anmen Hospital of China Academy of Chinese Medical Sciences

REFERENCES:
- [Background] Niccoli G, Montone RA, Lanza GA, Crea F. Angina after percutaneous coronary intervention: The need for precision medicine. Int J Cardiol. 2017 Dec 1;248:14-19. doi: 10.1016/j.ijcard.2017.07.105. Epub 2017 Aug 12. PMID 28807510
- [Background] Ambrose JA, Dangas G. Unstable angina: current concepts of pathogenesis and treatment. Arch Intern Med. 2000 Jan 10;160(1):25-37. doi: 10.1001/archinte.160.1.25. PMID 10632302
- [Background] Smith JN, Negrelli JM, Manek MB, Hawes EM, Viera AJ. Diagnosis and management of acute coronary syndrome: an evidence-based update. J Am Board Fam Med. 2015 Mar-Apr;28(2):283-93. doi: 10.3122/jabfm.2015.02.140189. PMID 25748771
- [Result] Jiang M, Zhang C, Zheng G, Guo H, Li L, Yang J, Lu C, Jia W, Lu A. Traditional chinese medicine zheng in the era of evidence-based medicine: a literature analysis. Evid Based Complement Alternat Med. 2012;2012:409568. doi: 10.1155/2012/409568. Epub 2012 Jun 6. PMID 22719784
- [Result] Zhang HJ, Wang ZX. Yin-yang and Zheng: Exported from Chinese medicine. Chin J Integr Med. 2014 Apr;20(4):250-5. doi: 10.1007/s11655-014-1777-z. Epub 2014 Apr 3. PMID 26972437
- [Derived] Tian PP, Wu QJ, Li J, Chen HW, Wu J, Deng YW, Xie ZC, Zhao W, Tan YQ. Efficacy and safety of Chinese herbal medicine Wen Xin granules for the treatment of unstable angina pectoris with Yang deficiency and blood stasis syndrome: study protocol for a randomized controlled trial. Trials. 2021 Nov 13;22(1):798. doi: 10.1186/s13063-021-05771-y. PMID 34774099